CLINICAL TRIAL: NCT06244121
Title: Effect of Pyridoxine as Add-on Therapy With Standard Treatment in Obsessive Compulsive Disorder Patients: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effect of Pyridoxine as Add-on Therapy in OCD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Sumaiya Nousheen Pinki, MD, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2023/7593
Record Dates: First submitted 2024-01-28; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: OCD
Keywords: Pyridoxine; OCD; RBC Glutathione; Plasma MDA; Vit B6
MeSH Terms: interventions — Pyridoxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (participant, investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment with pyridoxine (Experimental): This group will receive standard treatment with pyridoxine 25 mg twice daily for 8 weeks
  Interventions: Drug: Pyridoxine
- Standard treatment with placebo (Placebo Comparator): This group will receive standard treatment with placebo 25 mg twice daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridoxine — pyridoxine (Vitamin B6) will be given as an anti oxidant.
  Arms: Standard treatment with pyridoxine
Drug: Placebo — Placebo will be given in control group
  Arms: Standard treatment with placebo

SUMMARY:
Title:

Effect of Pyridoxine as Add-on Therapy with Standard Treatment in Obsessive Compulsive Disorder Patients: A Randomized, Double-Blind, Placebo-Controlled Trial

Purpose of the study:

This study aims to examine the effect of Pyridoxine with standard treatment in Obsessive Compulsive Disorder patients.

Method:

It will be a prospective type of interventional study to to assess the effects of Pyridoxine along with standard treatment in OCD patients. The study will be conducted in the Department of Pharmacology,BSMMU and Department of Psychiatry, BSMMU, from September 2022 to July 2024. A total of 76 OCD patients will be selected according to inclusion and exclusion criteria. The patients will be divided randomly into 2 groups: group A and group B. Group A will consist of 38 patients who will receive tablet pyridoxine 25 mg twice daily with standard treatment and group B would consist of 38 patients who will receive placebo twice daily along with standard treatment for 8 weeks. To see the effects of pyridoxine, Yale-Brown score of obsessive-compulsive disorders (Y-OCD) would be assessed by Yale-Brown Obsessive Compulsive Scale (Y-BOCS) at baseline (before pyridoxine administration) and 8 weeks after intervention(after pyridoxine administration). Biochemical parameters of oxidative stress markers such as plasma malondialdehyde (MDA), RBC glutathione (GSH) would be performed at baseline (before pyridoxine administration) and 8 weeks after intervention.

Ethical consideration:

The study will follow the principles of the Declaration of Helsinki and of the World Medical Assembly. Patients will be informed about the study in easy language and then informed consent will be taken. This study has no potential risk to the patients. Confidentiality will be strictly maintained.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is the fourth most common mental disorder in Bangladesh and around the world. Selective serotonin reuptake inhibitors (SSRIs) are commonly administered drugs for treating children and adolescents with OCD. The treatment of this condition has remained unsatisfactory, only 40-60% of patients with OCD respond to SSRIs, and about 40 to 60% of patients with OCD do not completely respond to this drug. Researchers throughout the world are involved to obtain new pharmacotherapy for the treatment of OCD. A good number of evidences have proved that oxidative stress plays a significant role in the pathophysiology of OCD.Researches so far have indicated that free radical induced injuries are involved in the pathology of OCD.Pyridoxine (Vit B6) is a water soluble vitamin, has anti oxidant effects.Therefore the present study has been designed to assess the effects of pyridoxine along with standard treatment upon OCD patients.

Aim: This proposed study is therefore an effort whether there is any role of Pyridoxine (vit B6) adjuncts with standard treatment produce better improvement than standard treatment alone in OCD patients. Method: This study will be a randomized, double-blind, placebo-controlled trial that will be conducted in the department of pharmacology, BSMMU in collaboration with the department of psychiatry, BSMMU, Dhaka from the day of approval by the IRB (Institutional Review Board) to July 2024. A total of 76 patients suffering from OCD will be selected according to inclusion and exclusion criteria. The diagnosis of patients suffering from OCD and the selection of drug and dosage would be performed by a senior professor of the psychiatry department. After completing the necessary formalities including informed consent of the patients, the patient would undergo a selected questionnaire Yale-Brown Obsessive Scale (Y-BOCS-10) to assess the severity of the disease. The patients would be randomly allocated into two arms: control and intervention. Patients in the intervention arm would consist of 38 patients who will receive standard treatment plus tab pyridoxine 25 mg twice daily for 8 weeks. On the other hand, the control arm would consist of 38 patients who will receive standard treatment plus a placebo for 8 weeks. The severity of symptoms will be assessed after 8 weeks follow-up. Biochemical parameters of oxidative stress markers (RBC glutathione, plasma MDA) will be measured at baseline and after 8 weeks.Along with the biochemical parameters, Yale-Brown score of obsessive-compulsive disorders (Y-OCD) would also be assessed by Yale-Brown Obsessive Compulsive Scale (Y-BOCS) at baseline and after 8 weeks. The regularity of medicine intake will be ensured over the telephone and from the patient's compliance sheet. Statistical analysis will be obtained by SPSS (statistical package for social science) version 24. The calculated 'p' value may suggest the level of significance (significant at p<0.05). Ethical consideration: After approval from IRB (Institutional Review Board) every eligible patient will be informed about the intervention and the study objectives. Patients will also be informed that they can participate or to withdraw at any time without compromising their medical care. Patient confidentiality will be strictly maintained. Patient's personal data regarding the name, age, sex, and other information will not be disclosed anywhere and will be used only for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with OCD diagnosed by Psychiatry Department of BSMMU.
* OCD patients fulfills Diagnostic criteria of DSM-5 (Diagnostic and Statistical Manual of Mental Disorders,5th Edition)

Exclusion Criteria:

* Patients with other psychological disorder
* Prior exposure to pyridoxine within last 2 months
* Pregnant and lactating mother
* Patients unwilling to participate or unwilling to give written consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
To examine the effect of Pyridoxine as add on therapy with standard treatment in Obsessive Compulsive Disorder patients. | 8 weeks
  To assess and compare the clinical improvement of OCD patients by Yale-Brown Obsessive Compulsive Scale (Y-BOCS),where minimum and maximum values are 0 (best) and 40 (worst) respectively, and compare plasma MDA in umol/L, RBC glutathione in mg/L levels at baseline and after 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sumaiya Nousheen, Dhaka, Bangladesh